CLINICAL TRIAL: NCT01334996
Title: Treatment of Systemic Mastocytosis With Tamoxifen
Brief Title: Use of Tamoxifen in Systemic Mastocytosis
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joseph Butterfield, PI, Mayo Clinic
Other Study IDs: 2506-04
Record Dates: First submitted 2007-12-25; First posted 2011-04-13 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Systemic Mastocytosis
MeSH Terms: conditions — Mastocytosis, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, the investigators will determine the utility of Tamoxifen, a non-cytotoxic agent, to improve quality of life, biochemical parameters, and bone marrow involvement in systemic mastocytosis patients having 1) up to 40% bone marrow infiltration by mast cells and/or 2) mediator-release symptoms which are not controlled by tolerated doses of standard "non-cytotoxic" medications regardless of the percentage bone marrow involvement by mastocytosis. The dose of Tamoxifen will be 40 mg/day and the duration of treatment will be for one year. Patients currently taking interferon alfa, imatinib mesylate, or cladribine will be excluded until these medications have been stopped.

DETAILED DESCRIPTION:
Not desired

ELIGIBILITY:
Inclusion Criteria:

* Systemic Mastocytosis

Exclusion Criteria:

* Current treatment with Imatinib mesylate, cladribine or interferon alpha.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic mastocytosis having up to 20% bone marrow involvement or clinical symptoms not controlled on current medications.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2005-02; Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Stability or reduction of the percent bone marrow involvement by mastocytosis, including stable mast cell morphology and phenotype. | 1 year
  up to 40% bone marrow infiltration by mast cells and/or 2) mediator-release symptoms which are not controlled by tolerated doses of standard "non-cytotoxic" medications regardless of the percentage bone marrow involvement by mastocytosis. The dose of Tamoxifen will be 40mg/day and the duration of treatment will be for one year.

SECONDARY OUTCOMES:
Stability or improvement in biochemical markers of systemic mastocytosis | 1 year
  Stability or improvement in biochemical markers of systemic mastocytosis (serum tryptase, calcitonin, urinary N-methyl histamine and prostaglandin F2 excretion/24 hours, liver function studies, lactic dehydrogenase, complete blood count with leukocyte differential)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph H Butterfield, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States